CLINICAL TRIAL: NCT01128647
Title: Disposal of Oral Fructose During Exercise
Status: Completed | Type: Observational
Sponsor: University of Lausanne (Other)
Responsible Party: Principal Investigator, Luc Tappy, MD, Professor of Physiology, University of Lausanne
Other Study IDs: Protocole 59/09
Record Dates: First submitted 2010-05-21; First posted 2010-05-24 (Estimated); Last update posted 2013-02-13 (Estimated); Status verified 2013-02

CONDITIONS: Carbohydrate Metabolism at Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Dietary Supplement: Fructose:glucose drink
Dietary Supplement: glucose drink

SUMMARY:
There is evidence that total carbohydrate oxidation during exercise is higher after ingestion of fructose:glucose mixture than after ingestion of equimolar amounts of glucose alone. This may possible contribute to improve performance, provided that the extra carbohydrate oxidation induced by fructose:glucose co-ingestion occurs in skeletal muscle. The present study aims at assessing the hypothesis that, during exercise, a substantial portion of oral fructose is converted into lactate prior to oxidation To identify the major pathways of fructose disposal, 7 healthy endurance trained male volunteers will be studied. For each participant the following measurement will be performed

* a measurement of maximal oxygen consumption (VO2 max) on an ergometric bicycle
* a 2 hour exercise protocol with oral administration of a glucose drink. 6,6-2H2 glucose (0.44 µmol/kg/min) and 13C3 lactate (2.25 µmol/kg/min) will be infused to calculate glucose and lactate kinetics. Indirect calorimetry will be performed to measure total carbohydrate oxidation and expired 13CO2 will be monitored to calculate whole body lactate oxidation
* a 2 hour exercise protocol with oral administration of a glucose:fructose (72 + 48 g every hour) mixture. 6,6-2H2 glucose (0.44 µmol/kg/min) and 13C3 lactate (2.25 µmol/kg/min) will be infused to calculate glucose and lactate kinetics. Indirect calorimetry will be performed to measure total carbohydrate oxidation and expired 13CO2 will be monitored to calculate whole body lactate oxidation
* a 2 hour exercise protocol with oral administration of a glucose:fructose (72 + 48 g every hour) mixture with fructose labelled with 13C6 fructose to evaluate exogenous fructose metabolic fate and oxidation. 6,6-2H2 glucose (0.44 µmol/kg/min) will be infused to calculate glucose kinetics. Fructose conversion into lactate and glucose will be evaluated by monitoring the systemic appearance of plasma 13C-labelled lactate and 13C-labelled glucose. Total exogenous fructose oxidation will be measured by monitoring 13CO2 production.

Based on these measurements, semi-quantitative estimates of total fructose oxidation, fructose conversion into glucose, fructose conversion into lactate, and oxidation of fructose-derived lactate will be obtained

ELIGIBILITY:
Inclusion Criteria:

* age between 18 and 35 years
* males
* good physical health
* weekly cycling training sessions (> 3 sessions/week)

Exclusion Criteria:

* diabetes or glucose intolerance
* past history of heart disease
* alcohol intake > 30 g/day
* smokers
* drug consumption

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy, endurance trained male volunteers
Sampling Method: Non-Probability Sample
Enrollment: 7 (Actual)
Dates: Start 2009-04; Primary Completion 2009-12 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Fructose conversion into lactate | during a 2 hour-exercise at 60% VO2 max

SECONDARY OUTCOMES:
Total exogenous fructose oxidation | during a 2 hour-exercise at 60% VO2 max
Fructose conversion into glucose | during a 2 hour-exercise at 60% VO2 max
Oxidation of lactate derived from fructose | during a 2 hour-exercise at 60% VO2 max

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Universitaire Vaudois, Lausanne, Switzerland

REFERENCES:
- [Derived] Lecoultre V, Benoit R, Carrel G, Schutz Y, Millet GP, Tappy L, Schneiter P. Fructose and glucose co-ingestion during prolonged exercise increases lactate and glucose fluxes and oxidation compared with an equimolar intake of glucose. Am J Clin Nutr. 2010 Nov;92(5):1071-9. doi: 10.3945/ajcn.2010.29566. Epub 2010 Sep 8. PMID 20826630